CLINICAL TRIAL: NCT00506870
Title: Economic and Medical Evaluation of Self-monitoring of Anticoagulation in a Population of Patients Recently Fitted With a Mechanical Heart Valve Compared to Conventional Anticoagulation Follow-up
Brief Title: Benefit of Self-monitoring of Anticoagulation Instrument
Acronym: 4A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry of Health, France (Other Government); Hoffmann-La Roche (Industry); Biodis (Unknown)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CHUBX2006/04; 2006/019
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-12

CONDITIONS: Mechanical Prosthetic Heart Valve Implantation; Patient Self Monitoring of Oral Anticoagulent Therapy
Keywords: Heart Valve Prosthesis Implantation; INR self monitoring; cost benefit evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Conventional follow-up of anticoagulation
  Interventions: Device: Conventional follow-up of anti-coagulation
- 2 (Experimental): Self-monitoring of anticoagulation
  Interventions: Device: INRatio / Coaguchek XS

INTERVENTIONS:
Device: INRatio / Coaguchek XS — INR measured by patient himself using INRation or Coaguchek device. And one follow-up of INR per month, measured in laboratory.
  Arms: 2
Device: Conventional follow-up of anti-coagulation — At least, one follow-up of INR per month. Measured in laboratory.
  Arms: 1

SUMMARY:
To evaluate the benefit economic and medical of self-monitoring of coagulation compared with conventional follow-up of anticoagulation in a population recently fitted with mechanical heart valves.

DETAILED DESCRIPTION:
Rationale/context:

Long term management of anticoagulant treatment is not straightforward, especially in patients bearing mechanical heart valves due to the requirement of maintaining a high INR over a narrow range.

Due to the narrow therapeutic window of AVK, undesirable events (hemorrhages, thromboembolic accidents) tend to be both serious and common leading to frequent admissions to hospital The self-monitoring of AVK, in addition to conventional monitoring of INR in the laboratory, is now being introduced in several countries (USA and Europe).

Main objective To evaluate the benefit economic and medical of self-monitoring of coagulation compared with conventional follow-up of anticoagulation in a population recently fitted with mechanical heart valves.

Secondary objectives

To compare over one year the effect of self-monitoring of coagulation with conventional follow-up of anticoagulation on:

* the impact of complications stemming from oral anticoagulant treatment (bleeding, thromboembolic episodes or death
* the proportion of monthly values of INR within the target range,
* the inherent cost of each strategy of monitoring of anticoagulation,
* the incidence of death, bleeding and thromboembolic episodes (each studied separately)
* The quality of life and the satisfaction of the patient To evaluate the patients' learning to be autonomous Diagram of the study Progress of the trial

A national, multicenter, randomized, blind trial, designed to examine the type of strategy used for monitoring anticoagulation in two parallel groups:

* a conventional follow-up of anticoagulation (monthly checks and adjustment of INR by the family doctor (GP))
* a self-measurement of anticoagulation by the patient at home using a Roche Diagnostics Laboratories test CoaguChek XS® or the Hemosense laboratories test INRatio® (weekly measurements and adjustment of INR by the family doctor) + a monthly laboratory check of INR

Inclusion criteria:

* adults (age ≥ 18 years), either sex
* patients fitted with one or more mechanical heart valves either alone or in combination with myocardial revascularization
* oral anticoagulant treatment
* patients with social security cover
* written informed consent signed by both patient and investigator Exclusion criteria
* women pregnant or liable to become pregnant during the study
* nursing women
* patients unable to master the self-monitoring procedures
* individuals under judicial control or enquiry
* patients consuming excessive amounts of alcohol ((>40g/j for men et >30g/j for women femmes ; 1 glass = 10g)
* patients on dialysis
* patients with incomplete understanding of instructions
* blind patients and those unable to read
* presence of circulating anticoagulant

Treatments/Strategies/Procedures:

1.1. Strategies of anticoagulation monitoring

After signature of informed consent and verification of criteria of eligibility, patients are randomly allocated into the following groups:

1.1.1. Conventional follow-up of anticoagulation In this group, the patients are instructed in the use of oral anticoagulants. INR is measured once a month in the laboratory. INR must lie in the therapeutic range designated by the investigative center as a function of the type and the location of the valve and any associated risk factors. If necessary, the family doctor adjusts INR on the day of the blood test and a new measurement is taken 48 hours later if dosage has been changed.

This algorithm is applied until the INR comes into the designated range.

1.1.2. Self-measurement of anticoagulation In this group, the patients are instructed in the use and monitoring of oral anticoagulants. They are further trained in the use of the self-monitoring test system.

Reference INR will be INR labo during first post operatives weeks up to the return at home because the self-measurement of anticoagulation maybe for lack of the fact of the anaemia, the inflammatory syndrome and the residues of heparin.

When the patients return at home, they take a measurement every week and if the result is abnormal, inform their family doctor. The INR must lie within the therapeutic range designated by the investigative center as a function of the type and the location of the valve and any associated risk factors. If necessary, the family doctor adjusts the INR on the same day as the self-measurement. A measurement is taken 48 hours later if the dosage has been changed.

This algorithm is applied until the INR comes into the designated range. INR is measured in the laboratory every month.

Main evaluation criteria:

Economic and medical evaluation of self-monitoring of coagulation compared with conventional follow-up of anticoagulation in a population recently fitted with mechanical heart valves.

Main secondary evaluation criteria:

* the impact of complications stemming from oral anticoagulant treatment (bleeding, thromboembolic episodes or death) within a population recently fitted with a mechanical hear valve.
* the proportion of monthly measurements of INR within the designated range,
* the inherent cost of each strategy of anticoagulation monitoring,
* the impact of death, bleeding and thromboembolic episodes (each studied separately),
* Evaluation of patients' learning of monitoring procedures.

Planned population size: 1050 patients, i.e.

* 350 in the group "Conventional follow-up of anticoagulation"
* 700 in the group "Self-measurement of anticoagulation" :

  * 350 using the Roche Diagnostics laboratories test CoaguChek XS®
  * 350 using the Hemosense laboratories test INRatio®

Time-line:

* Period of inclusion: 12-18 months
* Duration of participation by patients: 12 months
* Duration of trial: 30 months

ELIGIBILITY:
Inclusion Criteria:

* adults
* patients fitted with one or more mechanical heart valves either alone or in combination with myocardial revascularization
* oral anticoagulant treatment
* patients with social security cover
* written informed consent signed by both patient and investigator

Exclusion Criteria:

* women pregnant or liable to become pregnant during the study
* nursing women
* patients unable to master the self-monitoring procedures
* individuals under judicial control or enquiry
* patients consuming excessive amounts of alcohol ((>40g/j for men et >30g/j for women femmes ; 1 glass = 10g)
* patients on dialysis
* patients with incomplete understanding of instructions
* blind patients and those unable to read
* presence of circulating anticoagulant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 919 (Actual)
Dates: Start 2007-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Economic and medical evaluation of self-monitoring of coagulation compared with conventional follow-up of anticoagulation in a population recently fitted with mechanical heart valves. | 12 months

SECONDARY OUTCOMES:
- the impact of complications stemming from oral anticoagulant treatment (bleeding, thromboembolic episodes or death) within a population recently fitted with a mechanical hear valve. | 12 months
the proportion of monthly measurements of INR within the designated range | 12 months
the inherent cost of each strategy of anticoagulation monitoring | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Raymond ROUDAUT, Pr, Study Director — University Hospital, Bordeaux; Geneviève CHENE, Pr, Study Chair — University Hospital, Bordeaux; Raymond ROUDAUT, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Pôle Cardio-Thoracique - Hôpital Cardiologique du Haut-Lévêque - CHU de Bordeaux - Avenue de Magellan, Pessac, France